CLINICAL TRIAL: NCT02228954
Title: Watchful Waiting in Patients With Good and Intermediate Risk Metastatic Renal Cell Carcinoma; an Imaging Guided Observational Approach. Part of: Towards Patient Tailored Cancer Treatment Supported by Molecular Imaging. IMPACT Study: Imaging Patients for Cancer Drug Selection
Brief Title: IMaging PAtients for Cancer Drug selecTion - Renal Cell Carcinoma (IMPACT-RCC)
Acronym: IMPACT-RCC
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: IMPACT-RCC study
Record Dates: First submitted 2014-08-26; First posted 2014-08-29 (Estimated); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Clear-cell Metastatic Renal Cell Carcinoma; Kidney Neoplasms
Keywords: Clear-cell metastatic renal cell carcinoma; Positron-Emission Tomography
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Kidney Neoplasms | interventions — Molecular Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Renal Cell Cancer
  Interventions: Procedure: Molecular imaging

INTERVENTIONS:
Procedure: Molecular imaging

SUMMARY:
Rationale. In part of the patients with good and intermediate risk metastatic renal cell carcinoma (mRCC) the disease course is indolent and immediate start of systemic therapy is not necessary. By now, the investigators are not able to identify those patients with indolent disease and the minor group of patients with rapidly progressive disease. In patients with indolent disease, a watchful waiting period is preferred, since their quality of life will not be unnecessary hampered by adverse events and therapy resistance is not induced. This study aims to identify those patients for whom a watchful waiting period is possible by molecular imaging. Furthermore several types of systemic therapy are possible once the progression is proven. These systemic treatments are comparable in terms of efficacy, but not in terms of toxicity and their impact on quality of life. As a secondary objective, the usefulness of a decision aid guiding the choice of the patients is studied.

Objectives.

To assess in patients with good or intermediate prognosis mRCC who are eligible for watchful waiting, the added value beyond clinical work-up of:

1. FDG-PET and 89Zr-girentuximab-PET results measured at presentation to predict rapid progression (≤ 2 months after the baseline scan) under watchful waiting.
2. FDG-PET and 89Zr-girentuximab-PET results measured at presentation to predict prolonged indolent (≥12 months after the baseline scan) disease under watchful waiting.

To assess the value of a therapy choice decision aid for patients with progressive disease.

Study design. This is a multicenter non-blinded prospective observational study in 80 good and intermediate prognosis mRCC patients.

Study population. Patients with good or intermediate prognosis mRCC according to the Heng criteria, ≥18 years, without contra-indications for a watchful waiting period, able to provide informed consent.

Intervention. At baseline an FDG-PET-CT and 89Zr-girentuximab-PET will be made. During the watchful waiting period, disease evaluation by CT according to the RECIST criteria will be made frequently, until established progressive disease. At that moment, a second FDG-PET-CT and, in case of a positive 89Zr-girentuximab-PET-scan at baseline, a second 89Zr-girentuximab-PET will be performed and the decision aid is used to help the patient to choose their best treatment out of four options; pazopanib, sunitinib, combined interferon-α with bevacizumab and (only in case of a positive 89Zr-girentuximab-PET) radioimmunotherapy (RIT) with 177lutetium labelled girentuximab. Participation in the RIT trial is part of a separate phase II study.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness.

At baseline, a 18F-FDG-PET-CT and 89Zr-Girentuximab-PET will be performed. During the watchful waiting period CT's will be made. During therapy, follow-up will include standard laboratory analysis, and CT-scans on regular visits to the outpatient clinic. Side effects of the medication and adverse events as a consequence of the tumor biopsies may occur. The radiation exposure of both PET investigations is acceptable and requires no shielding after injection of 89Zr-labelled girentuximab. Patients may benefit from disease regression or stabilization. All three treatment choices has proven clinical benefit in this patient population. The risks of participation into the RIT trial are described in the phase II trial protocol, which already has been judged by the Medical Ethics Review Committee.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documented mRCC with a clear cell component
* Good or intermediate prognosis, defined as none (good risk) or 1-2 intermediate risk) of the below mentioned risk factors:

  * Karnofsky performance <80
  * Time from diagnosis detection of metastases < 1 year
  * Haemoglobin < lower limit of normal (LLN)
  * Corrected calcium > upper limit of normal (ULN)
  * Neutrophils > ULN
  * Platelets > ULN
* A watchful waiting period for 2 months is considered an option according to treating medical oncologist
* No prior systemic treatment for RCC (also non-adjuvant)
* Time from diagnosis of metastases < 3 months
* Able to provide written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Untreated central nervous system metastases, or symptomatic intracerebral metastases.
* Pregnant or breast feeding women.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that would make the subject inappropriate for study participation including any serious condition that could interfere with subject's safety, provision of informed consent, or compliance with study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with good or intermediate prognosis mccRCC according to the Heng criteria, ≥18 years, without contra-indications for a watchful waiting period, able to provide informed consent
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2021-10-19 (Actual)

PRIMARY OUTCOMES:
Time to progression | 1-5 years (End of study)
  To assess in patients with good or intermediate prognosis mRCC who are eligible for watchful waiting, the added value beyond clinical work-up of:
  1. FDG-PET and 89Zr-girentuximab-PET results measured at presentation to predict rapid progression (≤ 2 months after the baseline scan) under watchful waiting.
  2. FDG-PET and 89Zr-girentuximab-PET results measured at presentation to predict prolonged indolent (≥12 months after the baseline scan) disease under watchful waiting.

SECONDARY OUTCOMES:
Patient and physician questionnaires on the added value of the decision aid | 1-5 years (End of study)
  To assess the value of a therapy choice decision aid for patients with progressive disease

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - VU University Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Radboudumc, Nijmegen